CLINICAL TRIAL: NCT03158077
Title: Switching Strategy With Raltegravir + ABC / 3TC in Controlled HIV-1 Infection: Observational Retrospective Study at 48 Weeks - KIRAL Study
Brief Title: Switching Strategy With Raltegravir + ABC / 3TC in Controlled HIV-1 Infection
Acronym: KIRAL
Status: Completed | Type: Observational
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Other Study IDs: GeSIDA 8715
Record Dates: First submitted 2017-05-10; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Raltegravir + ABC/3TC: Switching or switching strategy with RAL and ABC / 3TC guidelines, 48 weeks before the start of the study

SUMMARY:
Retrospective observational study, multicentric with Spanish hospitals, in which a switching or change strategy with RAL and ABC / 3TC guidelines was used, in the48 weeks before the start of the study, in order to determine parameters of Effectiveness and security.

DETAILED DESCRIPTION:
The study consists of a 4-weeks data recording period, during which the follow-up information recorded by physicians in electronic or paper medical history will be analyzed from patients who opted for a change to that study pattern (RAL and ABC / 3TC).

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic infection with HIV-1.
* Patients older than 18 years.
* Patients in ART in whom RAL + ABC / 3TC has been initiated in at least 48 Weeks prior to the start of the study.
* To have used the RAL + ABC / 3TC as a switching or change strategy
* HIV virological control (CV ≤ 50 copies / ml) for at least 24 weeks prior to initiation of study regimen

Exclusion Criteria:

* NAIVE patients who have started treatment with this regimen
* Absence of digital or physical records of visits made for consultation
* Patients who underwent treatment change within 48 weeks prior to study initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients that initiated treatment with RAltegravis + ABC/3TC as a switching strategy
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Proportion of patients with undetectable viral load | 48 weeks
  Effectiveness in the virological control of RAL and ABC / 3TC

SECONDARY OUTCOMES:
Safety-changes in renal function: changes in creatinine values | 24 weeks following the change
Safety-changes in renal function: changes in glomerular filtration | 24 weeks following the change
Safety: Changes in serum levels of AST, ALT, FA, GGT and BIL | 24 weeks following the change
Safety: Changes in serum levels of AST, ALT, FA, GGT and BIL | 48 weeks following the change
Safety: Changes in serum cholesterol | 24 weeks following the change
  HDL and LDL cholesterol
Safety: Changes in serum triglycerides | 24 weeks following the change
Safety: Changes in serum cholesterol | 48 weeks following the change
  HDL and LDL cholesterol
Safety: Changes in serum triglycerides | 48 weeks following the change
Safety: Adverse events. | 24 weeks/48 weeks
  Frequency of adverse events
Safety:serious adverse events | 24 weeks/48 weeks
  Frequency of serious adverse events
Safety: frequency of adverse events leading to discontinuation of treatment. | 24 weeks/48 weeks
Safety: number of deaths | 24 weeks/48 weeks
Safety: frequency of laboratory abnormalities. | 24 weeks/48 weeks

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Hospital de Alicante, Alicante, Alcante
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Santa Lucia, Cartagena, Murcia
  - Hopital Severo Ochoa, Madrid
  - Hospital 12 de octubre, Madrid
  - Hospital Fundación Jimenez Díaz, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Prícipe de Asturias, Madrid
  - Hospital Ramón y cajal, Madrid
  - Hospital Univ. La Paz, Madrid
  - Complejo hospitalario de Toledo, Toledo
  - Hospital Rio Hortega, Valladolid
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No